CLINICAL TRIAL: NCT00518908
Title: Role of Volatile Anesthetics for Hepatic Protection in Ischemia-reperfusion: Postconditioning
Brief Title: Organ Protection With Sevoflurane Postconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: BECK SCHIMMER Beatrice, Professor, University Hospital Zurich, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StV 34-2007
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Hepatectomy
Keywords: Ischemia reperfusion injury; Organ protection
MeSH Terms: conditions — Reperfusion Injury | interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Sevoflurane for pharmacological postconditioning
  Interventions: Drug: Sevoflurane
- Propofol (Experimental): Anesthesia maintenance with propofol instead of Sevoflurane postconditioning
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — 3.2 Vol % for postconditioning

SUMMARY:
Organ protection, volatile anesthetics, postconditioning, hepatic surgery

DETAILED DESCRIPTION:
This study aims at the evaluation of a potential attenuation of ischemic-reperfusion injury in the liver with sevoflurane postconditioning upon reperfusion.

ELIGIBILITY:
Inclusion criteria:

* older than 18 years
* patients undergoing liver resection (benign or malignant tumors)

Exclusion criteria:

* non-german speakers
* laparoscopic liver resection
* coagulopathy (platelets < 50'000/ml, Quick < 50%)
* liver cirrhosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Liver transaminase AST | Postoperative phase until discharge
  Peak value

SECONDARY OUTCOMES:
ALT peak value | Postoperative phase until discharge
Course of transaminases | From the day before surgery, to 6 hours after surgery, up to postoperative day 7
Postoperative complications | Postoperative phase until discharge
Length of hospital stay | Postoperative phase until discharge
Need for prolonged intensive care unit stay (>24 hours) | Postoperative phase until discharge

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland